CLINICAL TRIAL: NCT01208961
Title: A Randomized, Open-label, Four-Way Crossover Study to Compare the Relative Bioavailability of a Single Dose of Epanova® With Lovaza® After a Low-Fat and High-Fat Meal
Brief Title: Epanova® Compared to Lovaza® In a Pharmacokinetic, Single-dose, Evaluation
Acronym: ECLIPSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Radiant Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OM-EPA-001
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Severe Hypertriglyceridemia
Keywords: Eicosapentaenoic Acid; Docosahexaenoic Acid; Hypertriglyceridemia; Omega-3 acid ethyl esters; Omega-3 carboxylic acids; Epanova; Lovaza; bioavailability; pharmacokinetics; low-fat meal; high-fat meal
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epanova-Lovaza-Epanova-Lovaza (Active Comparator)
  Interventions: Drug: Epanova (4 g) and Lovaza (4 g)
- Lovaza-Epanova-Lovaza-Epanova (Active Comparator)
  Interventions: Drug: Lovaza (4 g) and Epanova (4 g)

INTERVENTIONS:
Drug: Epanova (4 g) and Lovaza (4 g) — Single dose of Epanova (omefas), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Epanova (omefas), 4x1g capsules, taken with high-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters, 4x1g capsules, taken with high-fat meals
  Other Names: Note that omefas corresponds to omega-3 carboxylic acids
  Arms: Epanova-Lovaza-Epanova-Lovaza
Drug: Lovaza (4 g) and Epanova (4 g) — Single dose of Lovaza (omega-3-acid ethyl esters), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Epanova (omefas), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters,4x1g capsules, taken with high-fat meals, 7 day washout followed by single dose ofEpanova (omefas),4x1g capsules, taken with high-fat meals
  Other Names: Note that omefas corresponds to omega-3 carboxylic acids
  Arms: Lovaza-Epanova-Lovaza-Epanova

SUMMARY:
The objectives of this study are to compare the relative bioavailabilities of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in plasma from a single dose of Epanova or Lovaza during periods of high- and low -fat consumption.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged ≥18.
* Normal healthy volunteers based on medical history, clinical assessments, and laboratory assessments.
* Body mass index 25-35 kg/m2.
* Willingness to maintain current activity level.
* Willingness to adhere to the Therapeutic Lifestyle Changes (TLC)diet during screening and treatment washout periods.

Exclusion Criteria:

* Intolerance to omega-3 fatty acids, ethyl esters, or fish.
* Unable or unwilling to eat the study meals.
* Use of fish oil, other EPA or DHA containing supplements, or EPA and/or DHA fortified foods within 60 days of Visit 2, or during the study.
* Consumption of any fish within 7 days of Visit 2, or during the study.
* Use of flaxseed, perilla seed, hemp, spirulina, or black currant oils within 7 days of Visit 2, or during the study.
* History of malabsorption syndrome, Crohn's disease, acute or chronic pancreatitis, pancreatic insufficiency, small bowel resection.
* Women who are pregnant, lactating, or planning to become pregnant during the study period, or women of childbearing potential who are not using acceptable contraceptive methods. A woman is considered of childbearing potential if she is not surgically sterile or is less than 1 year since last menstrual period. Examples of acceptable contraceptive methods include abstinence, intrauterine device (IUD) or double barrier method, oral or injectable contraceptives.
* Recent history (past 12 months) of drug abuse or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
* Exposure to any investigational product, within 28 days prior to Visit 1.
* Any other condition the investigator believes would interfere with the subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Radiant Research, Chicago, Illinois, United States

REFERENCES:
- [Result] Davidson MH, Johnson J, Rooney MW, Kyle ML, Kling DF. A novel omega-3 free fatty acid formulation has dramatically improved bioavailability during a low-fat diet compared with omega-3-acid ethyl esters: the ECLIPSE (Epanova((R)) compared to Lovaza((R)) in a pharmacokinetic single-dose evaluation) study. J Clin Lipidol. 2012 Nov-Dec;6(6):573-84. doi: 10.1016/j.jacl.2012.01.002. Epub 2012 Jan 24. PMID 23312053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period started October 2010 and the last subject visit was November 2010. All subjects were qualified at the clinical site and eligibility was determined by the PI (one US clinical site).
Pre-assignment Details: This was a 4-way crossover study with a minimum 7-day washout period between each treatment. Subjects were healthy volunteers aged ≥ 18 with a body mass index 25-35 kg/m2 and who were not intolerant to omega-3 products or fish. Subjects were instructed to follow the TLC diet and abstain from omega-3 products or fish for screening and all periods.
Groups:
- Epanova-Lovaza-Epanova-Lovaza: Epanova (4 g) and Lovaza (4 g) : Single dose of Epanova (omefas; corresponds to omega-3 carboxylic acids), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Epanova (omefas), 4x1g capsules, taken with high-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters, 4x1g capsules, taken with high-fat meals
- Lovaza-Epanova-Lovaza-Epanova: Lovaza (4 g) and Epanova (4 g) : Single dose of Lovaza (omega-3-acid ethyl esters), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Epanova (omefas; corresponds to omega-3 carboxylic acids), 4x1g capsules, taken with low-fat meals, 7 day washout followed by single dose of Lovaza (omega-3-acid ethyl esters,4x1g capsules, taken with high-fat meals, 7 day washout followed by single dose of Epanova (omefas),4x1g capsules, taken with high-fat meals
Period: Low-Fat Period I
Arm/Group | Epanova-Lovaza-Epanova-Lovaza | Lovaza-Epanova-Lovaza-Epanova
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Low-Fat Period II
Arm/Group | Epanova-Lovaza-Epanova-Lovaza | Lovaza-Epanova-Lovaza-Epanova
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0
Period: High-Fat Period III
Arm/Group | Epanova-Lovaza-Epanova-Lovaza | Lovaza-Epanova-Lovaza-Epanova
Started | 26 | 26
Completed | 25 | 26
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: High-Fat Period IV
Arm/Group | Epanova-Lovaza-Epanova-Lovaza | Lovaza-Epanova-Lovaza-Epanova
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: To be included in the baseline analysis, subjects had to receive at least one dose of investigational product; all randomized subjects (n = 54) were included in the baseline analysis.
Groups:
- All Subjects: All subjects received both Epanova (E) and Lovaza (L), and both under fasted and fed conditions. Subjects were randomized 1:1 to one of the following treatment period sequences: ELEL or LELE.
Arm/Group | All Subjects
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-t): Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (the Final Time With a Concentration ≥ LOQ)
Description: Analyses of the outcome measures presented are for baseline-adjusted data for total (esterified and unesterfied) EPA and DHA since the presence of endogenous levels of these fatty acids would likely contribute to intra-subject variability and affect the analyses and interpretation.
Time Frame: Blood samples were obtained pre-dose at -1.0, -0.5, and 0 hours and after dose administration at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours.
Measure: Geometric Mean (Full Range); unit: nmol.h/mL
Groups:
- Epanova (Low-Fat Period): Single dose of Epanova (omefas), 4*1g capsules, taken after fasting 12 hours with no breakfast, followed with no-fat lunch and low-fat dinner
- Lovaza (Low-Fat Period): Single dose of Lovaza (omega-3-acid ethyl esters), 4*1g capsules, taken after fasting 12 hours with no breakfast, followed with no-fat lunch and low-fat dinner
Arm/Group | Epanova (Low-Fat Period) | Lovaza (Low-Fat Period)
Number analyzed (Participants) | 51 | 51
nmol.h/mL | 2650.1612 [689.2702 to 7883.4790] | 661.9490 [-603.7871 to 2967.3160]
Statistical Analysis 1: Comparison: Epanova (Low-Fat Period) vs Lovaza (Low-Fat Period); Results for the analyses of the High-Fat Periods were not posted because the critical comparison was the response of Lovaza versus Epanova to the clinically relevant low-fat diet to be used as adjunct in hypertriglyceridemia; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA on log-trans baseline-adj PK values using sequence, period, and treatments as fixed effects and subject nested within sequence as random effect; Ratio of Geometric Means = 400.36, 90% CI 2-sided [326.87 to 490.36]

2. Primary Outcome: AUC(Inf): Area Under the Plasma Concentration-time Curve From 0 to Infinity
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nmol.h/mL
Arm/Group | Epanova (Low-Fat Period) | Lovaza (Low-Fat Period)
Number analyzed (Participants) | 51 | 51
nmol.h/mL | 5219.56 [1388.8324 to 13802.1423] | 803.42 [217.7803 to 2810.6873]
Statistical Analysis 1: Comparison: Epanova (Low-Fat Period) vs Lovaza (Low-Fat Period); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, ANOVA — ANOVA model with baseline value as covariate, and treatment and user/non-user of lipid-altering drugs as factors. LSM estimate performed on log-scale; Ratio of Geometric Mans = 649.66, 90% CI 2-sided [511.75 to 824.75]

3. Primary Outcome: C(Max): Maximum Plasma Concentration
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nmol/mL
Arm/Group | Epanova (Low-Fat Period) | Lovaza (Low-Fat Period)
Number analyzed (Participants) | 51 | 51
nmol/mL | 225.7920 [38.7545 to 754.0992] | 61.0818 [21.0820 to 843.7832]
Statistical Analysis 1: Comparison: Epanova (Low-Fat Period) vs Lovaza (Low-Fat Period); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Ratio of Geometric Means = 369.66, 90% CI 2-sided [301.74 to 452.86]

ADVERSE EVENTS:
Description: The adverse event safety results were grouped and analyzed for the entire population since the OM-3 FFA and OM-3 EE treatments were single-dose administrations received by all subjects and the protocol was not developed as an exposure-response study design.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 28/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=54)
Diarrhoea (Infections and infestations) | 9 (10) — All events of diarrhea were considered mild, related to treatment, and had resolved during the trial.
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) — All events of hyperglycaemia were considered mild and not related to treatment. All events of hyperglycaemia except one were ongoing at the time of study completion.
Dizziness (Nervous system disorders) | 5 (5) — All events of dizziness were considered mild, related to treatment, and had resolved during the trial.
Headache (Nervous system disorders) | 10 (10) — Eight of the headache events were considered mild, related to treatment, and had resolved during the trial. Two headache events were considered mild, not related to treatment, and resolved during the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators may publish data arising from their own subjects. The PI will provide the Sponsor with copies of written publications (including abstracts and posters)at least 60 days in advance of submission. Data will be reviewed by all participating investigators prior to publication. The Sponsor will have 60 days to review all definitive publications, such as manuscripts and book chapters, and a minimum of 30 days to review all abstracts.